CLINICAL TRIAL: NCT01544933
Title: The Influence of the Ribs on the Gravity of Burst Thoracic Spine Fractures
Status: Completed | Type: Observational
Sponsor: Universidade de Passo Fundo (Other)
Responsible Party: Principal Investigator, Rodrigo Arnold Tisot, Principal investigator, Universidade de Passo Fundo
Other Study IDs: rtisot01
Record Dates: First submitted 2012-02-22; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2011-08

CONDITIONS: Burst Thoracic Spine Fractures
Keywords: spinal fractures; Thoracic vertebrae; spinal canal; kyphosis
MeSH Terms: conditions — Spinal Fractures; Kyphosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- burst fractures in vertebrae with true ribs: between T1 and T10
- burst fractures in vertebrae with floating ribs: between T11 and T12

SUMMARY:
The purpose of this study is to analyse the anatomic influence of the ribs related to the incidence and severity of burst spine fractures.

DETAILED DESCRIPTION:
To analyse the anatomic influence of the ribs related to the incidence and severity of burst spine fractures, with the measurements of kyphosis, vertebral collapse and vertebral canal narrowing

ELIGIBILITY:
Inclusion Criteria:

* burst fractures in thoracic spine

Exclusion Criteria:

* fractures that were not burst fractures in thoracic spine

Ages: 17 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with burst fractures of the thoracic spine treated by the Hospital Ortopedico de Passo Fundo
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
residual kyphosis | 3 years
  measurement of residual kyphosis by x-ray

SECONDARY OUTCOMES:
vertebral canal narrowing | 3 years
  vertebral canal narrowing in CT

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Tisot, Dr, Study Director — Hospital Ortopedico de Passo Fundo
Locations (1):
- Rodrigo Tisot, Passo Fundo, Rio Grande do Sul, Brazil